CLINICAL TRIAL: NCT04767958
Title: The RAPID COVID Study - Application of Point-of-Care COVID-19 Testing to Optimize Patient Care, Resource Allocation and Safety for Frontline Staff
Brief Title: The RAPID COVID Study - Application of Point-of-Care COVID-19 Testing
Acronym: RAPID COVID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device pulled from market due to inconsistent results.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20200858-01T
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a cohort study of participants falling into one of four groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients consulted upon by ICU, internal medicine, or cardiology for hospital admission (Experimental): All patients will have both standard care and point-of-care (experimental) NP swabs performed.
  Interventions: Diagnostic Test: Spartan COVID-19 Platform
- patients undergoing cardiac testing/procedures (Experimental): All patients will have both standard care and point-of-care (experimental) NP swabs performed.
  Interventions: Diagnostic Test: Spartan COVID-19 Platform
- patients awaiting surgery (Experimental): All patients will have both standard care and point-of-care (experimental) NP swabs performed.
  Interventions: Diagnostic Test: Spartan COVID-19 Platform
- Health Care Workers (Experimental): Health Care Workers who are being screened for COVID-19 will have both standard care and point-of-care NP swabs performed.
  Interventions: Diagnostic Test: Spartan COVID-19 Platform

INTERVENTIONS:
Diagnostic Test: Spartan COVID-19 Platform — Nasal-pharyngeal swab for testing on the Spartan Covid-19 platform

SUMMARY:
This study is being conducted to study the use and application of a point-of-care (POC) Covid-19 test developed by Spartan BioSciences and recently approved for clinical use by Health Canada.

DETAILED DESCRIPTION:
This RAPID COVID-19 study is a prospective, unblinded clinical trial. POC testing utilizing the Spartan Cube COVID-19 platform will be performed on a cohort of 2200 hospitalized patients who have been tested for COVID-19.

This cohort will be divided into three groups:

1. patients consulted upon by ICU, internal medicine, or cardiology for admission to the hospital
2. patients undergoing cardiac testing and/or procedures
3. patients awaiting surgery The results from the POC test will be compared to the results from the traditional hospital core lab test to determine sensitivity and specificity of the POC test.

An additional cohort of 500 quarantined health care workers will have the POC test performed and compared with the results from the traditional hospital core lab test.

ELIGIBILITY:
Inclusion Criteria:

* participants >/= 18 years of age
* patients for whom POC testing would change their course of treatment (in opinion of treatment team)

Exclusion Criteria:

* patients in whom conventional COVID-19 testing would not have otherwise been performed
* patients in whom immediate COVID-19 testing would not alter short-term treatment
* patients who refuse consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of POC testing as compared to core lab testing | 3 months
  Specificity, positive/negative predictive values will be derived

SECONDARY OUTCOMES:
Incidence in which decision making would have been altered by POC testing | 12 months
  examples include: ventilation decisions, use of ICU/isolation rooms, use of PPE, additional testing

OTHER OUTCOMES:
In hospital outcomes | 16 months
  In hospital outcomes include death, pneumonia, intubation, myocardial infarction, urgent revascularization,mechanical device support, transplant
Length of hospital admission | 16 months
  Total number of days in hospital will be collected

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No